CLINICAL TRIAL: NCT03323125
Title: Photoprotection Habits in Patients With Vitiligo
Acronym: VITISUN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17014J
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2017-10

CONDITIONS: Vitiligo; PHOTOPROTECTION; SUN-EXPOSITION; FITZPATRICK SCALE
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-Assessment Questionnaire — Self-assessment questionnaire with sun exposition, sun protection, vitiligo severity and vitiligo outbreaks, will be suggested to patient during medical consultation.

SUMMARY:
Intro:

Patients with vitiligo have a reduced protection on depigmented areas. To date, however, little is known about photoprotection habits in patients with vitiligo even though these patients are thought to have a decreased ability to efficiently protect their skin against sun damage. Moreover, exposure to artificial UV is one of the major elements of the treatment of vitiligo even though certain phenotypes of vitiligo could be photoinduced.

Hypothesis The Primary objective is to describe patients behaviour with sun exposition

The Secondary objectives are:

* to assess the link between sun exposition and vitiligo outbreaks
* to assess photoprotection habits according to initial phototype and vitiligo severity (SA-VES)
* To validate a short form of the VIPs questionnaire, a validated burden questionnaire.

Method We aim to conduct a prospective cross sectional study in patients with Vitiligo with the aim to evaluate sun protection habits in patients with vitiligo. For that purpose a semi-directed questionnaire to investigate the sun protection behavior of vitiligo patients (adults> 18 years of age) have been created by experts in the field. Vitiligo severity will be self-assessed by patients using a recently validated patient reported outcome, the SA-VES. Consecutive vitiligo patients consulting in the dermatology department of Henri Mondor Hospital (Créteil, France) will be proposed to participate the study after having given their oral consent. We are planning to enrol 500 patients.

In a first step, a descriptive analysis will be carried out in order to describe the characteristics of the sample. Basic summary statistics, such as proportions, means and standard deviations, will be used to characterize the population. In order to identify the factors associated with the severity of the disease on the one hand and the phototype on the other, comparisons between groups (severe versus non-severe and light phototype versus dark phototype) will be carried out by unconditional logistic regression. All potential predictors of severity will first be assessed individually, and Odds Ratio (OR), corresponding 95% CIs and P values will be calculated. The significance of the OR will be determined by the Wald test χ2, and the predictors with P <.20 will then be evaluated using a multivariate analysis with a pre-selection procedure. Possible interactions and multi-colinearity will be examined. Finally, the quality of fit of the final model will be evaluated using the logistic regression diagnostic procedure. P ≤ 0.05 will be considered as statistically significant. The Hosmer-Lemeshow test will be carried out to test the suitability of the model.

Conclusion This study will help to identify gaps in the knowledge of sun protection habits in patients with vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 y.o
* Men or women with Vitiligo

Exclusion Criteria:

* Oral or written opposition expressed by patient
* Patient under tutorship or curatorship
* cognitive dysfunction making communication or questionnaire filling impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to conduct a prospective cross sectional study in patients with Vitiligo (adults> 18 years of age). Consecutive vitiligo patients consulting in the dermatology department of Henri Mondor Hospital (Créteil, France) will be proposed to participate the study after having given their oral consent.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
estimation of skin sun reaction: Fitzpatrick scale | At inclusion
  Fitzpatrick scale is a numerical classification scale for human skin color that help to estimate skin reaction towards ultraviolet light exposure.
  It contains six categories, Type I is the fairest skin complexion and type VI is the darkest complexion :
  Type I (scores 0-6) always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II (scores 7-13) usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III (scores 14-20) sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV (scores 21-27) burns minimally, always tans well (moderate brown) Type V (scores 28-34) very rarely burns, tans very easily (dark brown) Type VI (scores 35-36) Never burns, never tans (deeply pigmented dark brown to darkest brown)

SECONDARY OUTCOMES:
vitiligo outbreak | At inclusion
  vitiligo outbreak: new stain in the 3 last months
Auto evaluation of vitiligo severity: SA-VES | At inclusion
  SA-VES (Self-Assessment - Vitiligo Extent Score)(1) is a patient reported outcome that measure the severity of vitiligo and its body extent from the patient perspective. Patients scored less than 10 are considered as less severe.
  (1)Development and validation of a patient-reported outcome measure in vitiligo: The Self Assessment Vitiligo Extent Score (SA-VES). van Geel N, Lommerts JE, Bekkenk MW, Prinsen CA, Eleftheriadou V, Taieb A, Picardo M, Ezzedine K, Wolkerstorfer A, Speeckaert R; international Vitiligo Score Working Group.. J Am Acad Dermatol. 2017 Mar;76(3):464-471.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION